CLINICAL TRIAL: NCT05015790
Title: Effect of VIrtual Reality Spectacles on the Management of Pain and Anxiety During the Insertion of the Implantable Catheter Chamber in the Operating Theatre in Cancer Patients
Brief Title: Effect of VIrtual Reality Spectacles on the Management of Pain and Anxiety
Acronym: LURVIDOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Valérie LOIZEAU, paramedical research coordination, Poissy-Saint Germain Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A00132-37
Record Dates: First submitted 2021-02-12; First posted 2021-08-20 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cancer
Keywords: Virtual reality, pain, cancer
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use of virtual reality Bliss Solution (Experimental): in the experimental arm the patient will receive the usual practice associated with a virtual reality session (20 minutes renewable) in a world chosen with the patient beforehand
  Interventions: Device: virtual reality Bliss Solution
- current practice, without Bliss Solution (No Intervention): patient will receive the usual practice, local anesthesia

INTERVENTIONS:
Device: virtual reality Bliss Solution — use virtual reality Bliss Solution
  Arms: use of virtual reality Bliss Solution

SUMMARY:
To assess the contribution of the use of virtual reality glasses on the pain perceived by patients during the installation of an ICP in the operating room under local anesthesia in the patient newly diagnosed with cancer

DETAILED DESCRIPTION:
The insertion of an implantable catheter chamber (ICH) is indicated in the case of prolonged or repeated infusions, particularly when the products injected are toxic to the venous walls, as is the case with cancer chemotherapy.

The insertion of a ICH is carried out in the operating theatre, usually under local anaesthesia. Although this operation is potentially painful and stressful, the question of its perception by the patient has not yet been addressed, nor the relevance of using non-invasive devices to alleviate the pain felt by the patient.

Among the proposals, virtual reality glasses Bliss Solution would be likely to improve patient management when a ICH is performed under local anaesthesia in the operating theatre.

The evaluation will be made on the contribution of the use of the Bliss Solution virtual reality glasses in the management of pain during the installation of an ICH under local anesthesia in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age
* Patient suffering from a cancerous pathology
* Patient taken care of for the installation of the ICH

Exclusion Criteria:

* Patient does not speak and understand French
* Patient who has had a previous ICH installation
* Patient with cognitive impairment
* Patient with pain perception disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-02-05 (Estimated); Study Completion 2022-06-05 (Estimated)

PRIMARY OUTCOMES:
The main assessment criterion is measured using the Visual Analogue Scale (VAS), which allows a self-assessment of the level of pain felt by the patient using a ruler rated from 1 to 10. | one year
  At the same the main evaluation criterion is a visual analogue scale (VAS) allowing a self-evaluation of the pain felt by the patient during the surgical intervention. The patient will rate their pain, on a scale from 0 for no pain to 10 for very severe pain. the data will be recorded at the time of the patient's installation, during the venipuncture and at the creation of the pocket.

SECONDARY OUTCOMES:
The evaluation criterion will be measured on the Hamilton scale measuring anxiety during an operation. | one year
  The anxiety felt by patients during the operation will be evaluated with the Hamilton Score.The Hamilton Depression Scale is a test for the intensity of anxiety and depressive disorders that can be used by everyone. It has 14 rated items from 0 to 3. The higher the score, the more severe the anxiety disorders. The minimum score is 0 and the maximum score is 42.

CONTACTS AND LOCATIONS:
Overall Officials: valerie M LOIZEAU, Principal Investigator — CHI Poissy
Locations (1):
- CH Poissy st Germain, Poissy, France

IPD SHARING:
Plan to Share IPD: No